CLINICAL TRIAL: NCT01236742
Title: Discontinuation of Orthokeratology on Eyeball Elongation (DOEE) Study. (1) Discontinuation of Lens Wear in Existing Ortho-k Children
Brief Title: Discontinuation of Orthokeratology on Eyeball Elongation in Myopic Children
Acronym: DOEE1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Menicon Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Pauline Cho, Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-ZG50-1
Record Dates: First submitted 2010-11-08; First posted 2010-11-09 (Estimated); Results first posted 2017-11-08 (Actual); Last update posted 2017-12-18 (Actual); Status verified 2017-11

CONDITIONS: Myopia
Keywords: children; corneal reshaping; myopia; myopia progression; orthokeratology
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- single-vision glasses and ortho-k lenses (Experimental): Children who are currently wearing ortho-k lenses at night for correction of refractive errors will be switched to wear single-vision glasses for the first 7 months and then switched back to ortho-k lenses for the next 7 months
  Interventions: Device: ortho-k lenses; Device: single-vision glasses
- ortho-k lenses (Active Comparator): Children who are currently wearing ortho-k lenses at night for the correction of refractive errors will continue with the current treatment and serve as the first control group
  Interventions: Device: ortho-k lenses
- single-vision glasses (Other): Children who are currently wearing single-vision spectacles in the daytime for correcting their refractive errors will continue with the current treatment and serve as the second control group
  Interventions: Device: single-vision glasses

INTERVENTIONS:
Device: ortho-k lenses — nightly wear of orthokeratology lenses to correct vision
  Other Names: orthokeratology; corneal reshaping therapy; Menicon Z Night lenses; Menicon Z Night Toric lenses
  Arms: ortho-k lenses; single-vision glasses and ortho-k lenses
Device: single-vision glasses — daily wear of spectacle glasses to correct vision
  Other Names: CR-39 lenses
  Arms: single-vision glasses; single-vision glasses and ortho-k lenses

SUMMARY:
The primary aim of this study is to compare eyeball elongation in existing ortho-k subjects who stop the treatment with subjects who continue ortho-k lens wear and control subjects wearing single-vision glasses.

DETAILED DESCRIPTION:
Children wearing ortho-k have been shown to have slower rate of myopic progression than those wearing single-vision spectacles (Cho et al. 2005) or soft lenses (Walline et al. 2009). Both studies showed that the effect of myopic control was most significant during the first six months of the treatment. It is unknown whether the myopic control effect would dissipate upon the discontinuation of the treatment or whether the myopic control effect only happened in the first six month of lens wear and was maintained thereafter. The current study aims at evaluating the effect of discontinuation of ortho-k treatment on myopic control in children who are currently on the treatment. This knowledge is necessary and important as patients/parents have concerns about the permanent dependency on ortho-k once they enrolled in the treatment.

Children who have been on the treatment for two years and have recently completed the myopic control studies at The Hong Kong Polytechnic University, i.e. the ROMIO, TO-SEE and HM-PRO studies, will be invited to participate in this 14-month study. Ortho-k subjects will be randomly assigned to study group or the ortho-k control group. The study group subjects will be required to stop lens wear for 7 months at the completion of the previous study (Phase I) and resume lens wear for next 7 months (Phase II). The ortho-k control group subjects will be required to continue the current treatment for another 14 months. Control subjects in the existing myopic control studies will be required to continue using the same treatment, i.e. single-vision glasses, for another 14 months. Rate of myopic progression among the 3 groups and at the two study phases will be determined and compared.

ELIGIBILITY:
Inclusion Criteria:

* Age 8-14 years old (inclusive)
* Subjects who have completed the ROMIO, TO-SEE or HM-PRO studies at The Hong Kong Polytechnic University
* Willingness to be randomized into groups (for ortho-k subjects)
* Availability for follow-up for at least 14 months

Exclusion Criteria:

* Non-compliance to the follow up schedule
* Non-compliance to the assigned optical correction (i.e. single-vision glasses or ortho-k lenses)
* Contraindication for contact lens wear and ortho-k (e.g. limbus to limbus corneal cylinder and dislocated corneal apex)
* Systemic or ocular) conditions which may affect contact lens wear (e.g. allergy and medication)
* Systemic or ocular conditions which may affect refractive development (e.g. Down syndrome, ptosis)

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 53 (Actual)
Dates: Start 2010-07; Primary Completion 2013-01 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pauline Cho, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- School of Optometry, The Hong Kong Polytechnic University, Hong Kong, Hong Kong, China

REFERENCES:
- [Background] Cho P, Cheung SW, Edwards M. The longitudinal orthokeratology research in children (LORIC) in Hong Kong: a pilot study on refractive changes and myopic control. Curr Eye Res. 2005 Jan;30(1):71-80. doi: 10.1080/02713680590907256. PMID 15875367
- [Background] Walline JJ, Jones LA, Sinnott LT. Corneal reshaping and myopia progression. Br J Ophthalmol. 2009 Sep;93(9):1181-5. doi: 10.1136/bjo.2008.151365. Epub 2009 May 4. PMID 19416935
- [Result] Cho P, Cheung SW. Discontinuation of orthokeratology on eyeball elongation (DOEE). Cont Lens Anterior Eye. 2017 Apr;40(2):82-87. doi: 10.1016/j.clae.2016.12.002. Epub 2016 Dec 27. PMID 28038841
- [Derived] Lawrenson JG, Shah R, Huntjens B, Downie LE, Virgili G, Dhakal R, Verkicharla PK, Li D, Mavi S, Kernohan A, Li T, Walline JJ. Interventions for myopia control in children: a living systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Feb 16;2(2):CD014758. doi: 10.1002/14651858.CD014758.pub2. PMID 36809645

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single-vision Glasses and Ortho-k Lenses | Ortho-k Lenses | Single-vision Glasses
Started | 18 | 19 | 16
Completed | 15 | 16 | 13
Not Completed | 3 | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Single-vision Glasses and Ortho-k Lenses | Ortho-k Lenses | Single-vision Glasses | Total
Number analyzed (Participants) | 18 | 19 | 16 | 53
Age, Continuous [Median (Full Range); unit: years] | 10 [10 to 14] | 11 [9 to 12] | 11 [9 to 13] | 11 [9 to 13]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 11 | 8 | 26
  Male | 11 | 8 | 8 | 27
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Chinese | 18 | 19 | 16 | 53
Region of Enrollment [Count of Participants; unit: Participants]
  China | 18 | 19 | 16 | 53
Axial length [Mean (Standard Deviation); unit: mm] | 24.83 (0.881) | 24.62 (0.772) | 24.72 (0.850) | 24.72 (0.823)

OUTCOME MEASURES:

1. Primary Outcome: Change in Axial Length
Description: To determine the changes in axial length in the first 7 months and the last 7 months in the three groups of subjects
Time Frame: Baseline, 7 months, and 14 months after baseline
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Single-vision Glasses and Ortho-k Lenses | Ortho-k Lenses | Single-vision Glasses
Number analyzed (Participants) | 15 | 16 | 13
mm
  Phase I (first 7 months) | 0.153 (0.021) | 0.087 (0.020) | 0.082 (0.022)
  Phase II (last 7 months) | 0.059 (0.014) | 0.068 (0.013) | 0.064 (0.015)

2. Secondary Outcome: Incidence of Adverse Effects
Description: The observation of serious and non-serious adverse events in the 14 months of study period
Time Frame: 14 months
Measure: Count of Participants; unit: Participants
Arm/Group | Single-vision Glasses and Ortho-k Lenses | Ortho-k Lenses | Single-vision Glasses
Number analyzed (Participants) | 18 | 19 | 16
Participants
  Serious adverse events | 0 | 0 | 0
  non-serious adverse events | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse effect data were collected within 2 months after completion of the study for subjects on ortho-k. The subjects were asked to return the contact lenses upon completion of the study and were dismissed once their refractive error and corneal shape were stabilized after cessation of ortho-k treatment. The time required was less than 2 months for all subjects.
Arm/Group | Single-vision Glasses and Ortho-k Lenses | Ortho-k Lenses | Single-vision Glasses
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/19 | 0/16
Other Adverse Events (participants affected / at risk) | 1/18 | 0/19 | 0/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single-vision Glasses and Ortho-k Lenses (N=18) | Ortho-k Lenses (N=19) | Single-vision Glasses (N=16)
Chalazion (Eye disorders) | 1 (1) | 0 (0) | 0 (0) — One subject in test group had to cease ortho-k lens wear due to chalazion in the left eye 2 months before the completion of study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No